**Study Title:** Cooking as Health Behavior in College Students

**NCT Number:** 00000397

Date: October 4, 2019



## **University of Vermont Consent to Participate in Research**

**Title of Research Project:** Examining Cooking as a Health Behavior in College Students

**Principal Investigator:** Lizzy Pope PhD, RD

**Sponsor:** University of Vermont, College of Agriculture and Life

Sciences; USDA Hatch Act Funds

#### Introduction

You are being invited to take part in this research study because you are a University of Vermont student and are interested in improving your cooking skills. This study is designed to investigate the role active cooking lessons and follow-up support may play in cooking behaviors and diet quality. This study is being conducted by the University of Vermont.

Your participation in this research study is optional. We encourage you to ask questions and take the opportunity to discuss the study with anybody you think can help you make this decision.

# Key Information to Help you Decide Whether or Not This Study is Right for You

- The study uses cooking classes, meal kits, and recipes to see if increasing someone's skill level and comfort with cooking can positively impact cooking frequency and diet quality.
- If you decide to participate in this study, you will be asked to choose whether you would like to:
  - Attend a hands-on cooking class for 6 weeks (2hrs each) OR
  - > Take part in no intervention during the Fall semester (other than data collection)
- Everyone who participates in the study (either classes or no classes) will be asked to:
  - Submit photos of a few meals eaten per week (10-15 min/week)
  - Report the number of meals you cooked each week (5-10 min/week)
  - Complete online questionnaires and 3 days of food tracking logs every 6 weeks (4x: ~2 hrs)
  - (Group dependent) Receive a meal kit delivery once per week (6 weeks)
  - (Group dependent) Receive emailed recipes once per week (6 weeks)
  - (only about 5 participants/group) Interview about meal photos (30 min)
- Total time commitment: 19 weeks (Oct 2019-April 2020); about 30 min-3 hrs/week (depending on group assignment and study phase).
- Risks: potential injuries during cooking exercises and possible breach of confidentiality

[Version 10/012019] 

 This study is designed to test whether cooking classes and follow-up intervention could improve someone's comfort with cooking and how often they cook.

The UNIVERSITY

Your participation is completely voluntary. The information above is only a brief summary of the study. If you are interested in learning more, it is important to read the following pages for additional detailed information about the study. If you decide to take part in the research, you will be asked to provide written consent at the end of this document.

We encourage you to ask questions and take the opportunity to discuss the study with anybody you think can help you make this decision.

# Why is This Research Study Being Conducted?

The purpose of this study is to determine if encouraging cooking as a health behavior actually improves health outcomes. Specifically, this study aims to understand if active cooking classes will increase cooking frequency and improve diet quality when compared with demonstration classes. If you think of cooking as a health behavior, cooking classes can be used like exercise classes. For someone trying to be more physically active, exercise classes give people the skills, social structure, and confidence to begin exercising on their own. We will also examine whether follow-up support in the form of meal kits and recipes increases cooking frequency and improves diet quality when compared with no follow-up support.

# **How Many People Will Take Part In The Study?**

Approximately 64 people will take part in this study.

# What Is Involved In The Study?

Participation requires a time commitment of 19 weeks over the course of the Fall and Spring semesters, 2019-2020. No study interventions or assessments will be scheduled during school breaks or holidays. Assessments in the form of questionnaires will be completed at the beginning of the study and the end of each study phase. The questionnaires will ask about your cooking behaviors, your cooking frequency, your eating and food behaviors, and an evaluation of the cooking class at the end of the study. The questionnaires should take approximately 30 minutes to complete. Additionally, participants will be asked to complete 3 days of tracking their diet using the Automated Self- Administered 24- Hour Dietary Assessment Tool (ASA-24). Each day of tracking using the tool should take less than 30 minutes. The data collected from the ASA-24 will be used by the study personnel to calculate a Healthy Eating Index score, which assess diet quality.

During a few cooking classes we will ask for volunteers to complete an interoceptive awareness evaluation. During this exercise, we will ask you to track your heartbeat for 30 seconds, and then tell us the result. Next, we will take your wrist pulse for 30 seconds. Results of this evaluation will then be compared with results from the Intuitive Eating Scale administered with


The UNIVERSITY the baseline survey set. Participation in the interoceptive awareness evaluation will be entirely voluntary, and all information collected will be kept confidential.

As part of the study, you will also be asked to take photos of a few meals you eat each week and submit these photos to the study staff. At the conclusion of the study, investigators will randomly select five participants from each group to interview about their photos. The interviews will ask questions about why the photos represented healthy or unhealthy meals to the participants, where the meals were prepared, how the photos may have changed over time, and how the various interventions may have affected the meals in the photos.

After initial assessments and tracking are complete, and should you choose to participate in this study, you will select whether you want to participate in the active cooking classes or control condition. Once enrolled in one of those categories you will be randomly assigned to one of two groups- one group will receive follow-up intervention (meal kits and recipes) and one group will receive no follow-up intervention. You will not be able to decide which group you are assigned to, and must be willing to be assigned to either group in order to participate.

Eligible participants who enroll in the cooking class intervention will be assigned to one of four scheduled class periods based on their stated availability. Once all classes are full (16 participants per class) a random assignment table will be used to determine whether each class group will receive follow-up intervention or no follow-up intervention. Participants not taking part in the cooking class intervention will be assigned at random to a group that will receive follow-up intervention or will not receive follow-up intervention. Participants will then be informed of their group assignment. Groups and participants will not be stratified by any criteria, and instead will be determined based upon participant availability.

All participants taking part in the cooking classes will attend six in-person cooking classes. These classes will take place every week at the scheduled time for six consecutive weeks. Classes will be two hours long and meet in the Foods Lab located in the Marsh Life Sciences building. Classes will be taught by a trained chef and all classes will follow the same recipe each week. Prior to the start of the cooking classes, every participant will take part in a Kitchen Intensive session at which the chef-instructor will introduce everyone to the kitchen space, review safety information, and demonstrate some of the skills and organization techniques that will be used during the classes. Participants will be given a brief lecture at the beginning of class that reviews the concepts of the week's recipe. Everyone will then work in teams of two to actively practice skills and cook the meal. All participants will receive the same printed information and also have an opportunity to sample the prepared food at the end of class. The lessons will be led by the same chef for all classes, will cover the same topics, and use the same recipes. All participants will be provided with the upcoming recipe and asked to prepare an organizational plan for preparing the recipe before coming to the weekly class meeting.

All participants enrolled in the control condition will not take part in any intervention during the Fall semester. Participants in the control condition will be asked to complete the same data


The UNIVERSITY measures as those in the cooking class intervention. These data measures include surveys and food logs. Participants will be offered gift cards and other giveaways for completing these data measures (see compensation section below).

Phase 2 of the study will begin after the start of the spring semester in mid-January. Two groups will begin receiving meal kit deliveries that include ingredients and instructions to make three meals designed to feed two people. All participants will be asked to complete data measures at the end of Phase 2 whether or not they were in a group that received meal kits.

Phase 3 of the study will begin after the end of Phase 2. The same participants who received meal kits will receive five healthy recipes designed by the study team that includes a chef and three registered dietitians. The recipes will be delivered by email at the beginning of the week for 6 weeks and will rely and build upon skills learned in the cooking classes. All participants will be asked to complete data measures at the end of Phase 3 whether or not they were in a group that received recipes.

### Outline of Groups and Study Phases

| Possible Group Assignments | | | |
|---|---|---|---|
| Group A | Active cooking classes followed by meal kits and recipes | | |
| Group B | Active cooking classes followed by no further instruction | | |
| Group C | Control Condition followed by meal kits and recipes | | |
| Group D | Control Condition followed by no further instruction | | |
| Study Phases | | | |
| Phase 1- Cooking classes | | Oct – Nov<br>2019 | All participants in active cooking classes will attend one kitchen intensive session followed by one cooking class per week for 6 weeks. |
| Data Collection | | Nov 2019 | Surveys, ASA-24 logs |
| Phase 2- Meal Kits | | Jan – Feb<br>2020 | Assigned participants will receive meal kit deliveries once per week for 6 weeks. |
| Data Collection | | Feb 2020 | Surveys, ASA-24 logs |
| Phase 3- Recipes | | March – April<br>2020 | Assigned participants will receive five healthy recipes by email once per week for 6 weeks. |
| Data Collection | | April 2020 | Surveys, ASA-24 logs |




### What Are The Benefits of Participating In The Study?

We hope that individuals who participate will learn the skills and behaviors necessary to help them cook healthy meals at home. However, you may or may not benefit from participating in this study as responses to cooking programs may vary from person to person. Everyone, however, will get expert information and feedback on cooking, meal planning, and choosing healthy foods. We expect that most participants will become familiar with at least some new kitchen equipment, cooking techniques, and/or ingredients over the duration of the study.

### What Are The Risks and Discomforts Of The Study?

There are minimal risks for participating in this study. If you are assigned to an active cooking class, you will be handling kitchen equipment including knives, blenders, and gas stoves. We will provide you with safety information and significant guidance before you use the equipment on your own. The chef-instructor and student assistants will always be present to ensure that you are using equipment safely. You will also be directed to safety procedures posted in the kitchen lab during the Kitchen Intensive session.

You may feel uneasy about answering the personal questions included in the interview. However, you do not have to answer any questions that make you feel uncomfortable. The information you provide will be kept confidential and not shared with non-research staff. No identifiable information about you will ever be published or shared without your consent.

## What Other Options Are There?

Community-based cooking classes are available through many local organizations including the University of Vermont Medical Center, Essex Resort, Healthy Living Market, City Market/ Onion River Co-op, Richmond Community Kitchen, and many others. Most classes are offered for a fee. The University of Vermont also offers cooking classes to university students. If you are a member of the WE Wellness Environment, you can participate in WEchopped. All students can sign up for Central Campus Dining Hall: Discovery Kitchen classes, once the semester calendar is available.

Home delivered meal kits are available through several companies for purchase. Meal kits can be ordered by number of meal per week and recipe amounts can be adjusted for household size.

#### **Are There Any Costs?**

There is no cost for participation other than your time. It will take you approximately 3 hours a week to attend the cooking classes and complete weekly data measures (photo uploads and cooking frequencies). It will take approximately 30 minutes to complete the online assessment questionnaires at the beginning and following each study phase, and approximately 90 total minutes to track food using the ASA-24 tool at each collection point.

#### What Is the Compensation?


In return for your time completing data measures, **All** study participants will be offered small gifts following each phase of the study. Gifts will be valued at \$5-\$25 and may include small kitchen equipment, gift cards, or cookbooks. Additionally, we will offer similar small incentives to encourage participants to submit the weekly photo uploads and weekly cooking frequencies.

# Can You Withdraw or Be Withdrawn From This Study?

You may choose to end your participation in the study at **any** time. Simply contact study personnel by phone (802-656-9526) or email (<u>malpaugh@uvm.edu</u>).

You may be asked to withdraw from the study if:

- You move more than 2 hours away from the University of Vermont during the study period.
- You sign up for meal delivery services outside of the study intervention.

Finally, the investigators reserve the right to end your participation in the research at any time.

## What About Confidentiality?

All the information you give us will be kept strictly confidential. You will be assigned identification numbers for the purposes of data collection and your name will not be connected to your ID numbers. A record of your progress will be kept in confidential form in the Marsh Life Sciences Building at the University of Vermont. Our study computers will require a password for access and any hard copies of data collection will be kept in a locked filing cabinet in a locked office.

Additionally, the results of this study may eventually be published and information may be exchanged between investigators; however, your confidentiality will be maintained during this process. Individual names and other personally identifiable information will not be used. The University of Vermont Institutional Review Board and regulatory authorities can be granted direct access to your original research records for verification of research procedures and/or data.

Please note that email communication is neither private nor secure. Though we are taking precautions to protect your privacy, you should be aware that information sent through e-mail could be read by a third party.

If you have questions or concerns about the use and disclosure of your health information, you should ask a member of the study team at insert phone number or the Chief Privacy Officer at The University of Vermont at (802) 656-2003.

#### **Contact Information**


You may contact Mattie Alpaugh the research coordinator at 802-656-9526 if you have any questions or concerns at any time before deciding to enroll in the study or during the course of the study. If you have any questions about your rights as a participant in a research project or for more information on how to proceed should you believe that you have been harmed as a result of your participation in this study you should contact the Director of the Research Protections Office at the University of Vermont at 802-656-5040.


#### STATEMENT OF CONSENT

You have been given and have read or have had read to you a summary of this research study. It has been explained to your full satisfaction. Should you have any further questions about the research, you realize you are free to contact the person conducting the study at the address and telephone number given below.

You understand the exact procedures you will undergo, including any potential benefits, risks, or discomforts.

You acknowledge that your participation is voluntary and are aware that you may refuse to participate or withdraw at any time without penalty or prejudice.

You understand that a record of your progress will be kept in confidential form in Marsh Life Sciences at the University of Vermont. You understand that the results of this study may eventually be published and that information may be exchanged between investigators, but that your confidentiality will be maintained.

You understand that you may contact the Director of the Research Protections Office at the University of Vermont (213 Waterman Building, 85 South Prospect Street; 656-5040) should you have any questions about your rights as a participant in a research study or for more information on how to proceed should you believe that you have been injured as a result of these research procedures.

You agree to participate in this study and you understand that you will receive a signed copy of this form.

| Signature of Subject | | <br>Date |
|----------------------------------------------------|------|-------------|
| Name of Subject Printed | | <br>Date |
| Signature of Principal Investigator or Designee | Date | |
| Name of Principal Investigator or Designee Printed | Date | <del></del> |

Principal Investigator: Lizzy Pope, PhD, RD

Address: Department of Nutrition and Food Sciences, 250 Carrigan Wing, UVM

Phone: 802-656-4262
